CLINICAL TRIAL: NCT03017794
Title: Evaluation of Neuroendocrine Differentiation as a Potential Mechanism of Tumor Recurrence Following Radiotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 16-008637
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Radiotherapy; Chromogranin A; Neuroendocrine differentiation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained for future research with permission of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gleason score 6 or less: Prostate adenocarcinoma with Gleason score 6 or less
- Gleason score 7: Prostate adenocarcinoma with Gleason score 7
- Gleason score 8 -10: Prostate adenocarcinoma with Gleason score 8 -10

SUMMARY:
This is a pilot study to test a hypothesis that a greater increase in serum chromogranin A (CgA) after a definitive radiotherapy (RT) with or without androgen deprivation therapy (ADT) is associated with a higher risk of prostate cancer recurrence after RT. Serum CgA level is measured before the start of RT and/or the start of neoadjuvant ADT for patients undergoing a definitive RT with or without ADT. CgA is also measured at various pre-defined post-RT time points. The study will analyze the followings: 1. Change in CgA level at various pre-defined post-RT time points from the baseline, 2. Correlation between the extent of post-therapy CgA change and Gleason score of malignancy, 3. Correlation between the extent of post-therapy CgA change and treatment outcome.

DETAILED DESCRIPTION:
Neuroendocrine differentiation (NED) in prostate cancer is a well-recognized phenotypic change by which prostate cancer cells transdifferentiate into neuroendocrine-like (NE-like) cells. Accumulated evidences have suggested that the prevalence of NE-like cells is associated with disease progression and poor prognosis.

NED can be induced by a therapeutic agent. Such therapeutic agents include RT and ADT. RT-induced NED represents a novel pathway by which prostate cancer cells survive radiotherapy and contribute to treatment failure and tumor recurrence. Chromogranin A is the serum biomarker for NED and correlates well with CgA-positive staining in biopsy specimens. It has been reported that elevated serum CgA is associated with poor therapeutic response, androgen-independent growth, and biochemical recurrence.

The study tests whether the extent of serum CgA increase by RT +/- ADT, which reflects radiation-induced NED, is correlated with the risk of prostate cancer recurrence following RT and a Gleason score of prostate carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Clinically localized prostate carcinoma, T1-T4 N0M0, any Gleason Score, any prostate-specific antigen (PSA), or Biochemical relapse with clinically suspicious (based on MRI or clinical examination) or biopsy-proven local recurrence in the prostatic fossa after a radical prostatectomy
* ≥18 years old
* Histologic diagnosis of prostate adenocarcinoma
* Signed informed consent

Exclusion Criteria:

* Biochemical relapse alone without clinically suspicious (i.e. no suspicious lesion on MRI of the prostatic bed) or biopsy-proven local recurrence in the prostatic fossa
* Regional pelvic node metastasis (N1)
* Distant metastasis (M1)
* Concurrent or previous cytotoxic medications
* Medical or psychological conditions that in the opinion of the investigator would not allow follow-up

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are to receive either definitive RT +/- ADT as a primary therapy or salvage RT +/- ADT as a salvage therapy for a biochemical relapse with local recurrence in the prostatic fossa following a radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-RT CgA and Gleason Score (GS) | 5 years 6 months
  Post-RT CgA will be correlated with Gleason score (GS).The Gleason score is calculated by adding together the two grades of cancer cells that make up the largest areas of the biopsied tissue sample. The Gleason score usually ranges from 6 to 10. The lower the Gleason score, the more the cancer cells look like normal cells and are likely to grow and spread slowly.
Chromogranin A (CgA) levels | 5 years 6 months
  Chromogranin A (CgA) levels will be recorded before radiation therapy (RT), during RT, and post-RT.

SECONDARY OUTCOMES:
Androgen deprivation therapy (ADT) and CgA | 5 years 6 months
  CgA levels of patients receiving RT plus androgen deprivation therapy (ADT) will be compared with CgA levels for patients receiving RT alone.
Post--therapy CgA in photon-based RT and proton-based RT | 5 years 6 months
  CgA levels in patients undergoing photon-based RT will be compared with CgA levels of those undergoing proton-based RT.
CgA and biochemical recurrence | 5 years 6 months
  CgA levels will be compared with biochemical recurrence of disease, defined as an increase in prostate-specific antigen (PSA) levels after treatment without other signs of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M. Phillips, MD, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials